CLINICAL TRIAL: NCT06098027
Title: [14C]CS0159 in Chinese Healthy Subjects for Mass Balance Phase I Study
Brief Title: Study of [14C]CS0159 in China Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cascade Pharmaceuticals, Inc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CS0159-001B
Record Dates: First submitted 2023-09-21; First posted 2023-10-24 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-10

CONDITIONS: Primary Biliary Cholangitis
MeSH Terms: conditions — Liver Cirrhosis, Biliary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]CS0159 (Experimental): Single oral dose of 4mg [14C]CS0159
  Interventions: Drug: [14C]CS0159

INTERVENTIONS:
Drug: [14C]CS0159 — Single oral administration of 4mg [14C]CS0159

SUMMARY:
Study of [14C]CS0159 in China Healthy Subjects.

DETAILED DESCRIPTION:
A phase I study to quantify the total mass balance in healthy subjects after a single dose of [14C]CS0159.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects between the ages of 18 and 45 years (inclusive).
2. Subjects should not weigh less than 50 kg, BMI between 19~26 kg/㎡.
3. No sperm donation or fertility plan during the study and within 12 months after the end of the study.
4. Understand the purpose and requirements of trial, subjects who have voluntarily participated in the study and signed the ICF, completion of tests as required.

Exclusion Criteria:

1. With abnormal and clinically significant comprehensive physical examinations, vital signs,laboratory examinations, 12-ECG, chest X-ray, and abdominal ultrasound.
2. 12-ECG QT(QTcF)>450ms.
3. The history of drug allergy.
4. Patients with malabsorption and gastrointestinal disorders or history of Vomiting, diarrhoea in the week prior to the screening period.
5. Patients with difficulty swallowing or interfere with drug absorption.
6. HBs Ag or E antigen, TPAb, or HIV-Ag/Ab positive person.
7. Have taken any clinical trial medication or participated in any other clinical trial within 3 months prior to the screening period.
8. Habitual constipation or diarrhoea.
9. Heavy smokers addicts
10. Heavy drinker addicts.
11. Has drug abuse history or positive drug abuse test results.
12. Heavy caffeine addicts.
13. Special dietary requirements.
14. Poor adherence or any other conditions judged by the investigator as not suitable for the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2023-10-23 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2023-11-02 (Actual)

PRIMARY OUTCOMES:
Mass Balance | Screening period (-48 hours) to 240 hours
  Mass balance recovery of total radioactivity in urine and fecal samples.
[14C] CS0159 metabolite | Screening period (-48 hours) to 240 hours
  Identification of the major metabolites of CS0159 in human plasma, urine and faeces, determine the main Determine the main biotransformation pathways and calculate the percentage of the administered dose of the prodrug and each metabolite in urine and faeces, and plasma prodrugs and circulating metabolites as a percentage of total exposure AUC.
Radioactivity of CS0159 | Up to 90 hours post dose
  Whole blood to plasma total radioactivity ratio
Area under the curve | Up to 90 hours post dose
  Total radioactivity in plasma PK: AUC
Highest radioactivity observed plasma concentration | Up to 90 hours post dose
  Total radioactivity in plasma PK: Cmax
Time for Cmax | Up to 90 hours post dose
  Total radioactivity in plasma PK: Tmax
Elimination half-life | Up to 90 hours post dose
  Total radioactivity in plasma PK: T1/2

SECONDARY OUTCOMES:
Blood plasma PK | Up to 90 hours post dose
  other major metabolites in plasma( if any).
Adverse events | Up to 240 hours post dose
  All subjects will be assessed for incidence and severity of adverse events (AEs) and serious AEs
AUC of CS0159 | Up to 90 hours post dose
  Area under the plasma concentration time curve of CS0159
Cmax of CS0159 | Up to 90 hours post dose
  Highest observed plasma concentration of CS0159
T1/2 of CS0159 | Up to 90 hours post dose
  Elimination half-life of CS0159
Tmax of CS0159 | Up to 90 hours post dose
  Time for Cmax of CS0159

CONTACTS AND LOCATIONS:
Overall Officials: Deng Rong, Study Director — Cascade Pharmaceuticals, Inc
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China